CLINICAL TRIAL: NCT00017511
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Cevimeline in the Treatment of Xerostomia Secondary to Radiation Therapy for Cancer in the Head and Neck Region
Brief Title: Cevimeline in Treating Patients With Dry Mouth Caused by Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000068698; DAIICHI-2011A-PRT003/004; UCLA-0104045
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Head and Neck Cancer; Oral Complications; Radiation Toxicity
Keywords: stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; oral complications; stage I squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage I verrucous carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II basal cell carcinoma of the lip; stage II verrucous carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage I squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; radiation toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — cevimeline

INTERVENTIONS:
Drug: cevimeline hydrochloride

SUMMARY:
RATIONALE: Cevimeline may be effective in treating dry mouth that is caused by radiation therapy for head and neck cancer. It is not yet known if cevimeline is more effective than no therapy in treating dry mouth caused by radiation therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of cevimeline in treating patients who have dryness of the mouth caused by radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of cevimeline vs placebo, in terms of dryness of the oral cavity and salivary flow, in patients with xerostomia secondary to radiotherapy for cancers in the head and neck region.
* Assess the safety of this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral cevimeline 3 times daily for 12 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo as in arm I.

PROJECTED ACCRUAL: A total of 280 patients (140 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Received more than 4,000 cGy of prior external beam radiotherapy for cancer in the head and neck region

  * Radiotherapy completed more than 4 months prior to study
* Clinically significant salivary gland dysfunction with grade 2 or 3 xerostomia
* At least 1 anatomically intact parotid gland
* No suspected or confirmed bilateral physical closure of salivary gland ducts
* No history of primary or secondary Sjogren's syndrome or other underlying systemic illness known to cause xerostomia independent of prior radiotherapy exposure

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%
* ECOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Hemoglobin at least 9.0 g/dL
* No anemia

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2 times ULN
* Lactate dehydrogenase no greater than 2 times ULN
* No evidence of active liver disease

Renal:

* Creatinine no greater than 2.5 mg/dL
* BUN no greater than 50 mg/dL
* No history of nephrolithiasis within the past 6 months

Cardiovascular:

* No history of significant cardiovascular disease
* No active congestive heart failure
* No uncontrolled angina
* No significant arrhythmia
* No myocardial infarction within the past 6 months

Pulmonary:

* No history of significant pulmonary disease
* No controlled or uncontrolled asthma
* No chronic bronchitis or chronic obstructive pulmonary disease that would limit avocational activities

Gastrointestinal:

* No history of significant gastrointestinal disorder
* No active pancreatic disease
* No gastroduodenal ulcers within the past 6 months
* No hypersensitive bowel conditions requiring pharmacologic therapy
* No inflammatory bowel disease
* No history of cholelithiasis within the past 6 months (unless cholecystectomy performed)

Other:

* No clinically significant laboratory abnormality
* No history of alcohol or drug abuse within the past 6 months that would preclude study
* No prior or concurrent acute iritis or narrow-angle (angle closure) glaucoma
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 30 days since other investigational new drug
* At least 4 weeks since prior systemic or ophthalmic pilocarpine
* No prior cevimeline
* No concurrent hyperbaric oxygen therapy
* No concurrent beta adrenergic antagonists, anticholinergic agents, cevimeline metabolism inhibitors, or other medications known to effect salivary function
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vitti, MD, Study Chair — Daiichi Sankyo
Locations (71):
- United States (71):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Cranial Pain Research, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Rebecca and John Moores UCSD Cancer Center, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Otolaryngology Associates, Colorado Springs, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Medical College of Georgia Hospital and Clinics, Augusta, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville, Kentucky
  - Tulane Cancer Center, New Orleans, Louisiana
  - Harbor Hospital Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Ear, Nose, and Throat Specialty Care of Minnesota, P.A., Minneapolis, Minnesota
  - University of Minnesota School of Dentistry, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Professional Otolaryngology Associates, Voorhees Township, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU - David B. Kriser Dental Center, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York at Stony Brook School of Medicine, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Gaston Memorial, Gastonia, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Clinical Research of Winston Salem, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oregon Cancer Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Head and Neck Associates, Havertown, Pennsylvania
  - Associated Otolaryngologist, Palmyra, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Eye and Ear Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Memorial Hospital Cancer Center - Chattanooga, Chattanooga, Tennessee
  - MultiSpecialty Clinical Research, Johnson City, Tennessee
  - Dial Research Associates, Inc., Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Dentistry, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Physicians Associates, PA, Laredo, Texas
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - McLean, Virginia
  - Seattle Institute for Biomedical and Clinical Research, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Southwest Washington Medical Center, Vancouver, Washington